CLINICAL TRIAL: NCT05817994
Title: Registry of Endoscopic Ultrasound Guided Assessment of the Liver (REGAL Study)
Brief Title: Endoscopic Ultrasound Guided Liver Biopsy and Portal Pressure Registry
Acronym: REGAL
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawn by the sponsor
Sponsor: Sheikh Shakhbout Medical City (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 313
Record Dates: First submitted 2023-03-18; First posted 2023-04-18 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2023-04

CONDITIONS: Liver Diseases; Liver Neoplasms; Liver Dysfunction; Liver Failure, Acute; Liver Fibrosis; Liver Inflammation
Keywords: liver; endoscopy; Biopsy; Ultrasound; EUS liver Biopsy
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms; Liver Failure, Acute; Liver Cirrhosis; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patient Registry aiming to provide regional evidence documenting the clinical merit of EUS (Endoscopic_ Ultrasound) guided liver biopsy, per local standard of practice, in patients with suspected liver disease indicated for an endoscopic intervention and a liver biopsy.

DETAILED DESCRIPTION:
The finding of this patient Registry may lead to recommendations towards optimizing liver biopsy procedures. If the study demonstrates the optimization of the number of interventions needed to reach diagnostic and therapeutic goals in the setting of suspected liver disease thanks to the utilization of Acquire compared to other liver biopsy procedures, this data can be used as part of economic messaging of the BSC Acquire Fine Needle Biopsy.

This Registry will document all relevant diagnostic and therapeutic radiologic - trans jugular or percutaneous - and endoscopic/endosonographic interventions which enrolled patients undergo when they are suspected to have liver disease and are indicated for an endoscopic procedure and liver biopsy. The study will help illustrate that an EUS guided approach for liver biopsy in patients with suspected liver disease that is indicated for:

Upper endoscopy and Liver biopsy will benefit both the patients and the hospitals from completing both procedures in one setting.

Where possible, the proposed Registry will also allow for the dynamic assessment of the severity of liver disease and for monitoring of changes to therapy for liver fibrosis and/ or portal hypertension. It is anticipated that the ability to monitor changes in liver status over time will become increasingly important as new therapies emerge in the field.

ELIGIBILITY:
Inclusion Criteria:

* Adult (per local age threshold)
* Suspected liver disease based on abnormal liver function tests, standard ultrasound, transient elastography (Fibro Scan) or CT or MRI of the liver
* Planned upper endoscopy to evaluate for varices
* Planned liver biopsy based on suspected hepatitis or cirrhosis

Exclusion Criteria:

* Severe Coagulation/bleeding disorder as defined by INR > 2 IU which cannot be corrected with FFP or Platelets < 50,000 per microliter which cannot be corrected with platelet transfusion.
* Severe organ failure considered unsafe to undergo sedation (ASA class 4 or 5)
* Inability to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll patients with suspected liver disease that are indicated for upper endoscopy for the assessment for esophageal varices and liver biopsy as per the local standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Number of endoscopic, endosonographic, and radiologic interventions undergone to reach a diagnostic liver biopsy [Phase 1] | 30 Days in Phase 1
  Number of endoscopic, endosonographic, and radiologic interventions undergone to reach a diagnostic liver biopsy in the setting of suspected liver disease from three months prior, to 30 days after the first upper Endoscopy procedure on study [ Phase 1]
Number of endoscopic, endosonographic, and radiologic interventions undergone to reach a diagnostic liver biopsy [Phase 2] | 12 months in phase 2
  Number of endoscopic, endosonographic, and radiologic interventions undergone to reach a diagnostic liver biopsy in the setting of suspected liver disease from three months prior, to 12 months after the first upper Endoscopy procedure on study [ Phase 2]

SECONDARY OUTCOMES:
Number of serious adverse events | 30 days (Phase 1), 12 months (Phase 2)
  Number of serious adverse events related to all livery biopsy study procedures (Phase 1 and Phase 2)
Number of Participants with Laboratory Abnormalities in Liver function Tests | from baseline to 6 months and from baseline to 12 months [Phase 2]
  number of participants with abnormal levels of liver function tests
Number of Participants with Noninvasive Liver Imaging abnormalities | from baseline to 6 months and from baseline to 12 months [Phase 2]
  number of participants with abnormal non-invasive liver imaging
Number of diagnostic liver biopsies | 13 months (phase 1 and 2)
  Number of diagnostic liver biopsies in radiologically guided compared to the EUS-guided liver.
  biopsy (Phase 1 and Phase 2)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asrani SK, Devarbhavi H, Eaton J, Kamath PS. Burden of liver diseases in the world. J Hepatol. 2019 Jan;70(1):151-171. doi: 10.1016/j.jhep.2018.09.014. Epub 2018 Sep 26. PMID 30266282
- [Background] Morales-Ruiz, Manuel, et al.
- [Background] Baran B, Kale S, Patil P, Kannadath B, Ramireddy S, Badillo R, DaVee RT, Thosani N. Endoscopic ultrasound-guided parenchymal liver biopsy: a systematic review and meta-analysis. Surg Endosc. 2021 Oct;35(10):5546-5557. doi: 10.1007/s00464-020-08053-x. Epub 2020 Oct 14. PMID 33052529
- [Background] Ali AH, Panchal S, Rao DS, Gan Y, Al-Juboori A, Samiullah S, Ibdah JA, Hammoud GM. The efficacy and safety of endoscopic ultrasound-guided liver biopsy versus percutaneous liver biopsy in patients with chronic liver disease: a retrospective single-center study. J Ultrasound. 2020 Jun;23(2):157-167. doi: 10.1007/s40477-020-00436-z. Epub 2020 Mar 5. PMID 32141043
- [Background] Bang JY, Ward TJ, Guirguis S, Krall K, Contreras F, Jhala N, Navaneethan U, Hawes RH, Varadarajulu S. Radiology-guided percutaneous approach is superior to EUS for performing liver biopsies. Gut. 2021 Dec;70(12):2224-2226. doi: 10.1136/gutjnl-2021-324495. Epub 2021 Mar 25. No abstract available. PMID 33766911
- [Background] ASGE Technology Committee; Trikudanathan G, Pannala R, Bhutani MS, Melson J, Navaneethan U, Parsi MA, Thosani N, Trindade AJ, Watson RR, Maple JT. EUS-guided portal vein interventions. Gastrointest Endosc. 2017 May;85(5):883-888. doi: 10.1016/j.gie.2017.02.019. Epub 2017 Mar 18. No abstract available. PMID 28320514
- [Background] Samarasena JB, Chang KJ. Endoscopic Ultrasound-Guided Portal Pressure Measurement and Interventions. Clin Endosc. 2018 May;51(3):222-228. doi: 10.5946/ce.2018.079. Epub 2018 May 31. PMID 29874904
- [Background] Huang JY, Samarasena JB, Tsujino T, Lee J, Hu KQ, McLaren CE, Chen WP, Chang KJ. EUS-guided portal pressure gradient measurement with a simple novel device: a human pilot study. Gastrointest Endosc. 2017 May;85(5):996-1001. doi: 10.1016/j.gie.2016.09.026. Epub 2016 Sep 29. PMID 27693644
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503